CLINICAL TRIAL: NCT00257400
Title: Interpersonal Psychotherapy for Depressed Women With Sexual Abuse Histories
Brief Title: Comparison of Two Psychotherapy Treatments for Depressed Women With a History of Sexual Abuse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH064528 (NIH); K23MH064528 (NIH); DSIR 8K-RTAT; NCT00843674 (obsolete NCT alias)
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: major depressive disorder; psychotherapy; childhood sexual abuse; trauma
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Wounds and Injuries | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal Psychotherapy (IPT) (Experimental): Interpersonal Psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy (IPT)
- Individual Psychotherapy (Active Comparator): Individual Psychotherapy
  Interventions: Behavioral: Individual Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy (IPT) — Interpersonal Psychotherapy
  Arms: Interpersonal Psychotherapy (IPT)
Behavioral: Individual Psychotherapy — Individual Psychotherapy
  Arms: Individual Psychotherapy

SUMMARY:
This study will compare the effectiveness of individual versus interpersonal psychotherapy in treating depressed women with a history of sexual abuse.

DETAILED DESCRIPTION:
Depression is a common but serious mental disorder that affects millions of people each year. Depression can severely impact people's lives, causing them to often feel sad and hopeless, as well as affecting people's sleep patterns, concentration, and energy levels. Women with a history of abuse are at an increased risk for developing symptoms of depression. However, treatments such as interpersonal psychotherapy and individual psychotherapy have been known to reduce symptoms of depression. This study will compare the effectiveness of individual and interpersonal psychotherapy in improving depressive symptoms and daily functioning in depressed women with a history of sexual abuse.

Participants in this study will undergo a two-part screening interview at the Strong Adult Ambulatory Clinic. This screening will include both written questionnaires and face-to-face interviews regarding any experiences of sexual or physical abuse; suicidal thoughts; family relationships; and current attitudes, thoughts, or feelings. Participants who meet all criteria will then be randomly assigned to receive one of two treatments: interpersonal psychotherapy or individual psychotherapy, which is considered usual care. All treatment sessions will be held at the Strong Adult Ambulatory Clinic. Participants assigned to receive interpersonal psychotherapy will attend weekly 50-minute sessions with a therapist. Interpersonal psychotherapy will focus on current interpersonal stressors in daily life, such as difficulties in close relationships or at work. Treatment will also help participants examine the relationship between their mood changes and interpersonal problems. Participants assigned to receive individual psychotherapy will undergo cognitive-behavioral therapy, supportive counseling, or a combination of the two. Participants will work with their therapists to decide upon a treatment plan designed to help changes in mood and other difficulties in daily life. The number and length of treatment sessions for this group will be determined on an individual basis. For all participants, evaluations consisting of questionnaires similar to those from the initial screening will be completed at mid-treatment, post-treatment, and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for unipolar major depressive disorder
* History of childhood sexual abuse before the age of 18
* Seeking outpatient psychotherapy treatment in a community mental health center

Exclusion Criteria:

* Meets DSM-IV criteria for major depression with psychotic features, bipolar disorder, schizophrenia, or mental retardation
* Active alcohol or substance abuse within 3 months of study entry date

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Measured at pre-treatment and Weeks 10, 24, and 36
Beck Depression Inventory | Measured at pre-treatment and Weeks 10, 24, and 36
Structured Clinical Interview for DSM-IV Diagnoses | Measured at pre-treatment and Weeks 10, 24, and 36

SECONDARY OUTCOMES:
Social Adjustment Scale | Measured at pre-treatment and Weeks 10, 24, and 36
Medical Outcomes Survey | Measured at pre-treatment and Weeks 10, 24, and 36
Post Traumatic Stress Disorder (PTSD) Symptom Scale | Measured at pre-treatment and Weeks 10, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Talbot, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Talbot NL, Conwell Y, O'Hara MW, Stuart S, Ward EA, Gamble SA, Watts A, Tu X. Interpersonal psychotherapy for depressed women with sexual abuse histories: a pilot study in a community mental health center. J Nerv Ment Dis. 2005 Dec;193(12):847-50. doi: 10.1097/01.nmd.0000188987.07734.22. PMID 16319710
- [Result] Talbot NL, Chaudron LH, Ward EA, Duberstein PR, Conwell Y, O'Hara MW, Tu X, Lu N, He H, Stuart S. A randomized effectiveness trial of interpersonal psychotherapy for depressed women with sexual abuse histories. Psychiatr Serv. 2011 Apr;62(4):374-80. doi: 10.1176/ps.62.4.pss6204_0374. PMID 21459988
- [Result] Smith PN, Gamble SA, Cort NA, Ward EA, He H, Talbot NL. Attachment and alliance in the treatment of depressed, sexually abused women. Depress Anxiety. 2012 Feb;29(2):123-30. doi: 10.1002/da.20913. Epub 2011 Nov 7. PMID 22065593
- [Result] Smith PN, Gamble SA, Cort NA, Ward EA, Conwell Y, Talbot NL. The relationships of attachment style and social maladjustment to death ideation in depressed women with a history of childhood sexual abuse. J Clin Psychol. 2012 Jan;68(1):78-87. doi: 10.1002/jclp.20852. Epub 2011 Nov 28. PMID 22125120
- [Result] Cankaya B, Talbot NL, Ward EA, Duberstein PR. Parental sexual abuse and suicidal behaviour among women with major depressive disorder. Can J Psychiatry. 2012 Jan;57(1):45-51. doi: 10.1177/070674371205700108. PMID 22296967
- [Result] You S, Talbot NL, He H, Conner KR. Emotions and suicidal ideation among depressed women with childhood sexual abuse histories. Suicide Life Threat Behav. 2012 Jun;42(3):244-54. doi: 10.1111/j.1943-278X.2012.00086.x. Epub 2012 Mar 12. PMID 22409700
- [Result] Cort NA, Gamble SA, Smith PN, Chaudron LH, Lu N, He H, Talbot NL. Predictors of treatment outcomes among depressed women with childhood sexual abuse histories. Depress Anxiety. 2012 Jun;29(6):479-86. doi: 10.1002/da.21942. Epub 2012 May 8. PMID 22570264